CLINICAL TRIAL: NCT06567730
Title: Comprehensive Comparison of Canine Retraction Using Nickel-titanium Closed-coil Springs Versus Elastomeric Power Chains During Orthodontic Treatment - A Split-mouth Randomized Controlled
Brief Title: Comparison of Canine Retraction Using Ni-ti Closed-coil Springs Vs Elastomeric Power Chains During Orthodontic Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Munnal Gulzar (Other)
Responsible Party: Sponsor-Investigator, Munnal Gulzar, Co-Investigator, Aga Khan University Hospital, Pakistan
Organization: Aga Khan University Hospital, Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-9110-28139
Record Dates: First submitted 2024-08-16; First posted 2024-08-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Root Resorption; Plaque Accumulation; Gingivitis
Keywords: canine retraction rate
MeSH Terms: conditions — Root Resorption; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ni-ti closed Coil spring (Experimental): For canine retraction, Ni-Ti closed-coil springs will be randomly allocated to the right and left quadrants of both arches
  Interventions: Other: Ni-ti Closed-coil Spring
- Elastomeric power chain (Active Comparator): For canine retraction, elastomeric power chains will be randomly allocated to the right and left quadrants of both arches
  Interventions: Other: Elastomeric Power chain

INTERVENTIONS:
Other: Ni-ti Closed-coil Spring — Ni-Ti closed-coil spring is a passive compressed spring made up of super elastic Nickel-titanium. Two eyelets are attached to each side of the coil to facilitate its application. The eyelets will be engaged in the hooks of the second premolar and canine brackets and will apply a force of 150 gm.
  Other Names: closing coil; closing coil spring
  Arms: Ni-ti closed Coil spring
Other: Elastomeric Power chain — Elastomeric power chains are resilient and latex-free orthodontic materials. They are made up of elastic material and consist of many connected rings. Each ring is engaged in a bracket to apply a force of 175-300 gm.
  Other Names: Power chain
  Arms: Elastomeric power chain

SUMMARY:
The objective of this study is to compare the canine retraction rate (in mm with a 100 mm marked scale) using Ni-Ti closed-coil springs versus elastomeric power chains during canine retraction in subjects with first premolar extractions over a period of three months.

After the extraction of all first premolars under local anesthesia. For canine retraction, Ni-Ti closed-coil springs and elastomeric power chains will be randomly allocated to the right and left quadrants of both arches.

Radiographic measurement (root resorption) and clinical measurements (canine retraction, plaque accumulation and gingival health) will be recorded at four points in time. First, at the start of the canine retraction (T0), after first month (T1), second month (T2) and third month follow-up (T3).

DETAILED DESCRIPTION:
RATIONALE:

Premolar extraction followed by canine retraction is one of the common practices in orthodontics to treat malocclusion such as severe crowding and proclination of anterior teeth. It is essential to know methods and techniques that result in minimum or no adverse effects on roots of teeth and periodontal health. This will help the clinicians to choose the best method that will result in a faster and more physiological closure of extraction spaces. Moreover, to the best of our knowledge, limited studies have compared the effects of Ni-Ti closed-coil springs and elastomeric power chains on canine root resorption, gingival health and plaque accumulation. It is necessary to establish a comparison between these methods, as it can help clinicians to provide better care and enhance the overall effectiveness of orthodontic treatment.

OBJECTIVE:

Primary Objective: The objective of this study is to compare the canine retraction rate (in mm with a 100 mm marked scale) using Ni-Ti closed-coil springs versus elastomeric power chains during canine retraction in subjects with first premolar extractions over a period of three months.

Secondary Objective: This study will also include an assessment of canine root resorption (in mm using periapical radiograph), dental plaque accumulation and gingival health (according to indices mentioned below with CPI-TN probe) using Ni-Ti closed-coil springs versus elastomeric power chains during canine retraction in subjects with first premolar extractions over a period of three months.

HYPOTHESIS:

Null Hypothesis: There is no significant difference between Ni-Ti closed-coil spring and elastomeric power chain on the canine root resorption, retraction rate, dental plaque accumulation and gingival health in subjects with first premolar extractions.

Alternate Hypothesis: There is a significant difference between Ni-Ti closed-coil spring and elastomeric power chain on the canine root resorption, retraction rate, dental plaque accumulation and gingival health in subjects with first premolar extractions.

DATA COLLECTION PROCEDURE:

After obtaining an approval from the Ethical Review Committee and taking informed consent and informed assent from the parents and child respectively, these patients will be recruited in the study as participants. Patients visiting the orthodontic clinic at the Aga Khan University Hospital Karachi will be included in this study. Detailed information regarding the study will be provided to the participants and they will be given the choice to either accept or refuse their inclusion in the study. After the extraction of all first premolars under local anesthesia, 0.018" stainless steel archwires will be inserted in the maxillary and mandibular arches. For canine retraction, Ni-Ti closed-coil springs and elastomeric power chains will be randomly allocated to the right and left quadrants of both arches. Radiographic measurement (root resorption) and clinical measurements (canine retraction, plaque accumulation and gingival health) will be recorded at four points in time. First, at the start of the canine retraction (T0), after first month (T1), second month (T2) and third month follow-up (T3). Canine retraction rate will be recorded by using a 100 mm marked scale. Data will be collected on an organized study proforma

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 13 - 40 years
* Patients undergoing fixed orthodontic treatment
* Patients requiring all first premolars extraction as part of orthodontic treatment
* Patients with all permanent teeth present and erupted (except for second and third molars)
* All patients who will sign the informed consent/assent form

Exclusion Criteria:

* • Patients with systemic diseases that can affect tooth movements

  * Patients with uncontrolled periodontal disease
  * Patients with craniofacial syndromes
  * Pregnant or lactating mothers
  * Patients with bracket failures greater than three times per bracket during the study
  * Patients on medications that can affect tooth movements
  * Patients with Nickel allergy

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Canine retraction rate | 3 months
  The retraction rate of canine will be the distance travelled divided by the time interval needed for closure of spaces. It will be noted at four-time intervals i.e at the start of the canine retraction (T0), after first month (T1), second month (T2) and third month follow-up (T3).

SECONDARY OUTCOMES:
Root resorption | 3 months
  Root resorption is a decrease in root length and width due to an inflammatory process. In orthodontics, during tooth movement, areas of necrosis develop called hyalinized areas, which result in root resorption. Periapical radiographs will be taken to assess the amount of root resorption by determining the length of the tooth from the cusp tip to the root apex
Gingival health | 3 months
  Gingival index is a grading system that is used to assess the health of the gingiva. It consists of four grades including, Grade 0, 1, 2 and 3. The increase in grade indicates the compromised gingival health of the teeth.
Plaque index | 3 months
  Plaque index is a grading system used to assess the amount of plaque present at the gingival margins and helps in assessing oral health. It consists of four grades including, Grade 0, 1, 2 and 3. The increase in grade indicates the increased amount of plaque along the gingiva.

CONTACTS AND LOCATIONS:
Overall Officials: Mubassar Fida, BDS,FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wazwaz F, Seehra J, Carpenter GH, Papageorgiou SN, Cobourne MT. Duration of canine retraction with fixed appliances: A systematic review and meta-analysis. Am J Orthod Dentofacial Orthop. 2023 Feb;163(2):154-172. doi: 10.1016/j.ajodo.2022.08.009. Epub 2022 Dec 1. PMID 36464569
- [Background] Kulshrestha RS, Tandon R, Chandra P. Canine retraction: A systematic review of different methods used. J Orthod Sci. 2015 Jan-Mar;4(1):1-8. doi: 10.4103/2278-0203.149608. PMID 25657985
- [Background] Makhlouf M, Aboul-Ezz A, Fayed MS, Hafez H. Evaluating the Amount of Tooth Movement and Root Resorption during Canine Retraction with Friction versus Frictionless Mechanics Using Cone Beam Computed Tomography. Open Access Maced J Med Sci. 2018 Feb 5;6(2):384-388. doi: 10.3889/oamjms.2018.066. eCollection 2018 Feb 15. PMID 29531610

DOCUMENTS (1):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT06567730/Prot_000.pdf